CLINICAL TRIAL: NCT06369896
Title: The Usefulness of Disposable Digital Single-operator Cholangioscopy and Intraductal Ultrasound in the Assessment of Nonicteric Biliary Strictures: A Prospective Observational Study
Brief Title: Digital Single-operator Cholangioscopy and Intraductal Ultrasound for Nonicteric Biliary Strictures
Acronym: Spy+IDUS
Status: Not yet recruiting | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jong Ho Moon, Professor Jong Ho Moon, Soonchunhyang University Hospital
Other Study IDs: SpyIDUSForNonictericStricture
Record Dates: First submitted 2024-01-21; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cholangiocarcinoma; Biliary Stricture
Keywords: intraductal ultrasound; digital single-operator cholangioscopy; indeterminate biliary stricture
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nonicteric stricture cohort: Patients with nonicteric biliary stricture

SUMMARY:
This study aims to evaluate the usefulness of disposable digital single-operator cholangioscopy (SOC) and intraductal ultrasound (IDUS) for the accurate diagnosis of indeterminate biliary stricture.

DETAILED DESCRIPTION:
Although early and accurate diagnosis of cholangiocarcinoma from the biliary stricture is important, accurate differential diagnosis is still difficult even in computed tomography and magnetic resonance imaging. We planned to evaluate the usefulness of disposable digital single-operator cholangioscopy (SOC) and intraductal ultrasound (IDUS) for the accurate diagnosis of biliary stricture.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 19 to under 80
2. Presence of nonicteric biliary stricture
3. Previous endoscopic sphincterotomy or papillary balloon dilatation

Exclusion Criteria:

1. Bleeding tendency (INR > 1.5 or platelets < 50000 mm3)
2. Contraindication to ERCP

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with indeterminate nonicteric (Bilirubin < 2mg/dL) biliary stricture
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-05-05 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of SOC | From enrollment through study completion, an average of 1 year
  sensitivity, specificity, and accuracy of SOC

SECONDARY OUTCOMES:
Diagnostic accuracy of IDUS | From enrollment through study completion, an average of 1 year
  sensitivity, specificity, and accuracy of IDUS
Technical success of SOC | From the time the cholangioscope is inserted into the working channel of the endoscope until it is removed
  Successful observation of extrahepatic duct using SOC
Technical success of IDUS | From the time the intraductal probe is inserted into the working channel of the endoscope until it is removed
  Successful observation of extrahepatic duct using IDUS
Adverse event | From enrollment through study completion, an average of 1 year
  All adverse event according to the American Society of Gastrointestinal Endoscopy criteria

IPD SHARING:
Plan to Share IPD: Undecided